CLINICAL TRIAL: NCT02735486
Title: Randomized, Controlled Trial of Ginger Extract Consumption for Healthy Males at Risk of Developing Cardiovascular Disease
Brief Title: Acute Effects of Ginger Extract Consumption on Risk Markers of Cardiovascular Disease
Acronym: G-CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PHYTOVAS II
Record Dates: First submitted 2015-12-08; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Disease
Keywords: Ginger; blood pressure; flow mediated dilatation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginger drink (Experimental): Experimental: Ginger drink (300 ml) to be consumed during the study visit
  Interventions: Dietary Supplement: Ginger drink
- Placebo: Super pure water (Placebo Comparator): Super Pure water low in nitrate content
  Interventions: Dietary Supplement: Placebo: Super pure water

INTERVENTIONS:
Dietary Supplement: Ginger drink — 300 ml ginger drink
  Arms: Ginger drink
Dietary Supplement: Placebo: Super pure water — Placebo: Super pure water
  Arms: Placebo: Super pure water

SUMMARY:
The primary aim of the study was to investigate the acute effect of ginger drink consumption on the risk markers of cardiovascular disease.

DETAILED DESCRIPTION:
A randomized, single-blind human intervention study involving 22 healthy male volunteers was designed to investigate the acute effects of ginger drink consumption on risk markers of cardiovascular disease (CVD). The primary outcome measure is reduction in blood pressure while the secondary outcome measures are improvement in flow mediated dilatation (FMD) and changes in plasma biochemical profile parameters related to CVD. Participants were given 300 ml of ginger extract or water (placebo) with breakfast, followed by a lunch at 2 hours on two visits separated by 2 weeks. Blood and urine samples were collected at regular intervals as well as blood pressure measurement done during the two visits. Vascular function was measured by flow mediated dilatation (FMD) and pulse wave velocity (PWV) at baseline, 2 and 4 hours after the the consumption of the study drink and placebo. The blood and urine samples were analysed for changes in lipid profile and other markers of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy males,
* Age (30 - 65) years,
* Not diabetic or plasma glucose > 7 or on anti-diabetic drugs and not on anti- hypertensive drugs.
* Subjects < 10% risk of cardiovascular disease

Exclusion Criteria:

* Women,
* Men younger than 30 years and older that 65 years,
* Men who are sick or on anti-diabetic and anti-hypertensive drugs.
* Men who have history of heart attack or stroke within the last 12 months
* Men who are on lipids lowering drugs

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Reduction in blood pressure (BP) | Six (6) hours
  Reduction in blood pressure (BP)

SECONDARY OUTCOMES:
Flow mediated dilatation | Six (6) hours
  Improvement in vascular function measured as percentage (%) increase in FMD

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy PE Spencer, Professor, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No